CLINICAL TRIAL: NCT01750398
Title: A Phase II Study of Bipolar Androgen-based Therapy for Men With Androgen Ablation NaÃ-ve Recurrent Prostate Cancer
Brief Title: Bipolar Androgen-based Therapy for Prostate Cancer (BAT)
Acronym: BAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1298; NA_00077460 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Prostate Cancer
Keywords: Testosterone, Leuprolide, Goserelin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; Testosterone; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADT plus IV testosterone (Experimental): Men with castration-resistant prostate cancer will initiate androgen deprivation therapy (ADT) with an LHRH agonist (e.g. goserelin or leuprolide) for a total of 6 months. After this initial "lead-in" castration phase, patients will receive intermittent intramuscular testosterone cypionate or testosterone enanthate (T) at a dose of 400 mg while continuing on ADT.
  Interventions: Drug: Testosterone cypionate; Drug: Goserelin; Drug: Leuprolide

INTERVENTIONS:
Drug: Testosterone cypionate — DEPO-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. DEPO-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
  Other Names: Testosterone
Drug: Goserelin — Goserelin is a hormone therapy, for intramuscular injectionis. It is classified as an "LHRH agonist."
  Other Names: Zoladex
Drug: Leuprolide — Leuprolide is a gonadotropin-releasing hormone (GnRH) agonist. For intramuscular injection.
  Other Names: Lupron Depot

SUMMARY:
The purpose of this study is to determine the safety and clinical effects of alternating androgen deprivation therapy with testosterone therapy in men with recurrent prostate cancer as first line hormonal therapy, to assess the effect of alternating therapy on quality of life and metabolic changes associated with androgen-deprivation therapy.

DETAILED DESCRIPTION:
This is an open-label, single site, single arm pilot study designed to determine the efficacy and safety of alternating androgen deprivation therapy (ADT) and parenteral testosterone in men with recurrent or newly metastatic prostate cancer. Eligible patients will initiate ADT with Luteinizing hormone-releasing hormone (LHRH) agonist (e.g. goserelin or leuprolide) if not surgically castrated for a total of 6 months. After this initial 6 month lead-in phase, patients will continue on ADT every three months but will also receive an intramuscular gluteal injection with either testosterone cypionate or testosterone enanthanate (T) at a dose of 400 mg every 4 weeks for a total of 3 injections (i.e.12 weeks of therapy).Both formulations of T have identical pharmacokinetics; exhibiting the same serum testosterone profile after intramuscular injection into healthy volunteers. Patients will then cycle back to ADT only for 12 weeks. This route and dose of T was selected based on data demonstrating that it produces an initial supraphysiologic serum level of testosterone (i.e. > 3-8 times normal level) with eugonadal levels achieved at the end of two weeks and return to low serum T levels by the fourth week post-injection. The investigators have termed this rapid cycling between supraphysiologic to low/castrate serum T Bipolar Androgen-based Therapy (BAT). One BAT cycle will be defined as 24 weeks (i.e. 12 weeks on T; 12 weeks off T). Patients will receive two cycles (i.e. 48 weeks) of BAT in total (see Study Scheme below). Upon completion of the 18 month study period patients will be assessed for response and will then have the option to continue on intermittent or continuous ADT at the discretion of their treating physician.

Patients will have prostate specific antigen (PSA) and imaging studies during the screening period. A second set of studies will be performed at the end of the 6-month LHRH agonist therapy lead-in period. Based on prior studies the investigators expect >80% of patients to have a PSA <4 ng/ml and without evidence of PSA progression after 6 months of ADT (Hussain et al. 2006; Crook et al. 2012). At the end of the lead-in phase only patients who either achieve a ≥50% reduction in PSA from their screening baseline (i.e. a major PSA response) or have a PSA < 4 ng/ml and are without signs of progression will be allowed to continue on the study. All others will be removed from study and replaced. Those replaced individuals will be considered to have not met the primary endpoint in our final analysis. PSA progression will be assessed at the end of the 18 month study period. Standard Prostate Cancer Working Group 2 (PCWG2) criteria for PSA progression will be used (Scher et al. 2008).

The primary endpoint for this trial will be the percent subjects with a PSA <4 ng/ml and without PSA progression at the end of the 18 month treatment period. Secondary endpoints will include: the rate of progression based on imaging and clinical assessments, percent of patient who have a complete PSA response (PSA < 0.2 ng/ml), metabolic changes, changes in quality of life as assessed through standard questionnaires, and safety.

CT and bone scans will be performed at the end of the second full cycle of BAT (i.e. at the end of the 18 month study period) and be used to assess for radiographic progression. Soft tissue metastasis will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (v1.1). Bone metastasis will be evaluated per the standard PCWG2 criteria. This requires the appearance of at least 2 new lesions with a confirmatory bone scan. For patients demonstrating radiographic progression the investigators will require a confirmatory scan after an additional 8 weeks so as not to misconstrue a tumor flare with true disease progression. A subject will be considered to have clinically progressed if he develops pain that, in the opinion of the investigator, is secondary to his cancer; he develops a pathologic fracture or other skeletal event. If there is uncertainty regarding whether a symptom is due to a patient's cancer, the subsequent workup will be at the investigator's discretion. Of the endpoints, only clinical progression will result in early study termination.

To evaluate the effect BAT has on the metabolic syndrome associated with ADT the investigators will monitor a number of parameters at baseline prior to initiation of ADT, after 6 month "Lead-in" phase of ADT and after the 2nd cycle of T. Studies will include measurements of bone density,estradiol, sex hormone binding globulins, fasting lipids, metabolic parameters (insulin, fasting glucose, hemoglobin A1c, leptin, TSH, T3, fibrinogen, C-reactive protein, serum C-telopeptide, blood pressure, Body Mass Index (BMI), body weight). Quality of life (QOL) will be recorded through a series of questionnaires. These surveys include the RAND-SF36 Quality of Life Survey, the Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P), the International Index of Erectile Function (IIEF), the International Prostate Symptom Score (IPSS) and a visual pain scale. Each of these instruments has been previously validated and is used extensively in clinical trials to assess the effects of treatment intervention on quality of life. QOL will be assessed at screening, after Lead-In Phase and at the end of each cycle of T or ADT.

Additional plasma and serum samples will be drawn and banked at -80°C at baseline prior to initiation of ADT, prior to initiating a cycle of T or ADT and upon completion of the study. These samples will be used for biologic and immunologic correlates. Examples of studies that may be performed include, but are not limited to: quantitative immunoglobulins, T-cell receptor excision circles (TREC) levels and circulating DNA studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Performance status ≤2.
3. Documented histologically confirmed adenocarcinoma of the prostate.
4. No prior AD therapy (i.e. surgical castration LHRH agonist, LHRH antagonist) as treatment for recurrent or metastatic disease (may have received neoadjuvant, concurrent and/or adjuvant AD therapy in the context of definitive local therapy if it was administered ≥ 1 year prior to recurrence).
5. No prior treatment with second line hormonal therapies (flutamide, bicalutamide, nilutamide, ketoconazole, abiraterone acetate or MDV3100) is permitted.
6. Prior treatment with 5-alpha reductase inhibitors (e.g. finasteride or dutasteride) for treatment of benign prostatic hyperplasia (BPH) is permitted, but patients must be off therapy for ≥ 6 months prior to enrolling on study
7. No prior treatment with chemotherapeutic regimens allowed.
8. Prior treatment with non-hormonal investigational agents is permitted.
9. Evidence of rising PSA on two successive dates > 2 weeks apart. There is no maximum or minimum PSA requirement to come on study.
10. Patients must have ≤ 10 total sites of bone metastases and no evidence for lung or liver or other parenchymal metastases documented within 28 days of enrollment on trial
11. Patient may have lymph node metastases with no single lymph node >5 cm short axis diameter
12. Patients must be asymptomatic with no sites of pain due to prostate cancer.

Exclusion Criteria:

1. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
2. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
3. Evidence of disease that, in the opinion of the investigator, would put the patient at risk from testosterone therapy (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction).
4. Requires urinary catheterization for voiding as a result of tumor obstructing the urinary outflow tract; catheterization is permitted if due to a non-oncologic cause (e.g urethral stricture or atonic bladder).
5. No prior history of deep venous thrombosis or pulmonary embolism within 5 years prior to enrollment in the study
6. Abnormal liver function (bilirubin, AST, ALT ≥ 3 x upper limit of normal)
7. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
8. Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within 5 years prior to enrollment in the study
9. Inability to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denmeade S, Lim SJ, Isaaccson Velho P, Wang H. PSA provocation by bipolar androgen therapy may predict duration of response to first-line androgen deprivation: Updated results from the BATMAN study. Prostate. 2022 Dec;82(16):1529-1536. doi: 10.1002/pros.24426. Epub 2022 Aug 8. PMID 35938545

RESULTS

PARTICIPANT FLOW:
Groups:
- ADT Plus IM Testosterone: Men with castration-resistant prostate cancer will initiate androgen deprivation therapy (ADT) with an LHRH agonist (e.g. goserelin or leuprolide) for a total of 6 months. After this initial "lead-in" castration phase, patients will receive intermittent intramuscular testosterone cypionate or testosterone enanthate (T) at a dose of 400 mg while continuing on ADT.
  Testosterone cypionate: DEPO-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. DEPO-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate.
  Goserelin: Goserelin is a hormone therapy, for intramuscular injectionis. It is classified as an "LHRH agonist."
  Leuprolide: Leuprolide is a gonadotropin-releasing hormone (GnRH) agonist. For intramuscular injection.
Period: ADT Lead In Phase
Arm/Group | ADT Plus IM Testosterone
Started | 33
Completed | 29
Not Completed | 4
Period: Bipolar Androgen Thearpy Phase
Arm/Group | ADT Plus IM Testosterone
Started | 29
Completed | 26
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 63 [46 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
PSA [Median (Full Range); unit: ng/mL] | 27.6 [5.6 to 257.3]
PSA doubling time [Median (Full Range); unit: months] | 5 [1 to 23]
Gleason score (higher score is associated with worse outcomes) [Number; unit: Number of patients] — Gleason score was based on clinical interpretation of the needle biopsy specimen or prostatectomy specimen by an expert pathologist. A pathologist examined this tissue specimens under the microscope and assigned a Gleason score based on the microscopic appearance of the prostate cancer.
  Number of patients
    Gleason 6 | 3
    Gleason 7 | 16
    Gleason 8 | 5
    Gleason 9 | 9
Local treatment [Number; unit: Number of patients]
  No local treatment | 3
  Radiation | 8
  Radical prostatectomy | 22
ECOG [Number; unit: Number of patients] — ECOG 0: no functional limitation.
  ECOG 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Determination of ECOG score was based on clinical assessment.
  Number of patients
    ECOG 0 | 31
    ECOG 1 | 2
Any metastatic disease [Number; unit: Number of patients]
  Positive for metastases | 20
  No metastases | 13
Patients with bone metastases [Number; unit: Number of patients]
  No bone metastases | 19
  Positive for bone metastases | 14
Patients with RECIST evaluable disease [Number; unit: Number of patients]
  No RECIST evaluable lesions | 20
  Positive for RECIST evaluable lesions | 13

OUTCOME MEASURES:

1. Primary Outcome: Patients With PSA <4 ng/mL at the End of the Study
Description: To determine the clinical effects of BAT in men with recurrent prostate cancer as first line therapy. This will be accomplished by assessing the number of patients achieving a PSA <4 ng/ml at the end of the trial.
Time Frame: 18 months
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 29
participants | 17 [12 to 21]

2. Secondary Outcome: Radiographic or Clinical Progression
Description: To evaluate the number of men treated per the bipolar androgen therapy phase of the trial who developed radiographic or clinical progression. Radiographic progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Clinical progression was defined as new symptoms that can be attributed to progressive prostate cancer (e.g. new/worsening pain, urinary obstruction, cord compression, bone fractures).
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 29
participants
  Patients with radiographic/clinical progression | 6
  Patients without radiographic/clinical progression | 23

3. Secondary Outcome: Complete PSA Response
Description: To evaluate the number of patients who achieve a complete PSA response (i.e. serum PSA <0.2 ng/ml) at the end of the study
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 29
participants
  Patients with PSA <0.2 ng/ml | 3
  Patients with PSA ≥0.2 ng/ml | 26

4. Secondary Outcome: Change in C-telopeptides
Description: Change in c-telopeptides following Round 1 of BAT (9 months) compared to the timepoint immediately following the ADT Lead-In (6 months)
Time Frame: 6 months and 9 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 33
pg/ml | -159.77 (190.66)

5. Secondary Outcome: Quality of Life Survey
Description: To measure quality of life through the RAND-SF36 (short-form 36 questionnaire) Quality of Life Survey, the Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P), the International Index of Erectile Function (IIEF), the International Prostate Symptom Score (IPSS) and a visual pain scale. Note that for all scales, higher scores indicate better quality of life/function, with the exception being the visual pain scale, where a higher score indicates more pain.
  RAND-SF36: SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Range is from 0 to 100.
  FACT-P: A tool used for assessing the health-related quality of life in men with prostate cancer. Range is from 0 to 156.
  IIEF: Is a measure of erectile function. Range is from 5 to 25. IPSS: A tool used to measure symptoms related to prostatic disease. Range is from 0 to 35.
  Visual pain scale: A tool used to track pain level. Range is from 0 to 10.
Time Frame: 3 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 33
units on a scale
  Change in SF-36 after round 1 of BAT | 3.2 [-20 to 48]
  Change in FACT-P after round 1 of BAT | 3.5 [-30 to 50]
  Change in IIEF after round 1 of BAT | 10 [-4 to 59]
  Change in IPSS after round 1 of BAT | 0 [-9 to 8]

6. Secondary Outcome: Change in Weight
Description: Change in weight is measured from baseline to 6 months (i.e. following ADT lead in) and from 6 months to 9 months (i.e. from post-ADT to the end of cycle 1 of BAT).
Time Frame: Baseline, 6 months and 9 months.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 33
kg
  Following ADT lead in | 2.08 (4.99)
  Following round 1 of BAT | 1.21 (1.99)

7. Secondary Outcome: Change in Waist Circumference
Time Frame: Bseline, 6 months and 9 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ADT Plus IM Testosterone
Number analyzed (Participants) | 33
cm
  Following ADT lead in | 3.9 (11.7)
  Following round 1 of BAT | -1.09 (1.54)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | ADT Plus IM Testosterone
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 23/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADT Plus IM Testosterone (N=29)
Hot flashes (Endocrine disorders) | 15
Edema (Blood and lymphatic system disorders) | 11
Weight gain (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 3
Pain (General disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Mood changes (Psychiatric disorders) | 1
Loss of libido (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Palpitations (Cardiac disorders) | 1
Facial flushing (Skin and subcutaneous tissue disorders) | 1
Dyspnea with exertion (Respiratory, thoracic and mediastinal disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No